CLINICAL TRIAL: NCT02008903
Title: Phase 2 Study of Esophageal String Test in Diagnosing Eosinophilic Esophagitis
Brief Title: Esophageal String Test in Eosinophilic Esophagitis
Status: Active, not recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: University of Illinois at Chicago (Other); Northwestern University (Other); OSF Healthcare System (Other)
Responsible Party: Sponsor
Other Study IDs: 07-0223; FD-R-G04086-01 (Other: FDA)
Record Dates: First submitted 2013-12-06; First posted 2013-12-11 (Estimated); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Eosinophilic Esophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- EoE active disease: Inflammation as defined by >15 eos / HPF
- EoE remission: No inflammation in EoE patients after treatment
- normal control: No inflammation

SUMMARY:
The overall goal of this study is to develop a novel minimally invasive device, the Esophageal String Test (EST) to monitor esophageal inflammation during treatment of the rare disease Eosinophilic Esophagitis (EoE) in a safe and efficacious manner.

This study is broken down into 2 specific aims:

Specific Aim 1: Identify the EoE Biomarker Panel (EBP) that will improve the sensitivity and specificity of the EST for documenting esophageal inflammation in a 1-hour time point.

Specific Aim 2: Validate the ability of the EST EBP to monitor therapeutic efficacy in a 1-hour sampling time.

Funding Source - FDA OOPD

DETAILED DESCRIPTION:
Eosinophilic esophagitis (EoE) is an increasingly recognized rare disease of children and adults characterized by symptoms including nausea, vomiting, abdominal pain, dysphagia and food impaction that occur in conjunction with esophageal eosinophilia. To date, the only method to make EoE diagnoses and follow treatment responses in EoE is invasive endoscopy with biopsy. While endoscopy is generally safe, an accurate, less invasive, inexpensive, comprehensive and durable test is urgently needed to determine therapeutic efficacy. To address this need, the investigators will use a novel application of an existing technology, the Enterotest™ (a string-based test used to detect intestinal Giardiasis), to measure esophageal inflammation (herein termed the Esophageal String Test - EST). The investigators supportive Preliminary Data provide proof-of-principle for the ability of ESTs to capture esophageal inflammatory mediators in luminal samples from patients affected with EoE. The investigators prospective study demonstrates that: (1) levels of eosinophil-derived granule proteins (MBP1, EDN, ECP, EPX, CLC/Gal-10) in esophageal mucosal biopsies correlate with levels quantitated in EST-captured samples, i.e., levels in luminal secretions captured by the EST correlate with mucosal inflammation, and (2) these luminal biomarkers of eosinophilic inflammation significantly correlate with EoE disease activity. These findings provide strong support for using ESTs as novel minimally invasive instruments to monitor therapeutic efficacy in EoE. The global objective of this project is therefore to bring the "Esophageal String Test" (EST) to commercialization, so that it can be used to monitor therapeutic efficacy in children and adults with EoE. The investigators hypothesize that ESTs will capture an EoE Biomarker Panel (EBP) reflective of disease activity. The Specific Aims are to: (1) Identify an EoE Biomarker Panel (EBP) that will improve the sensitivity and specificity of the EST for monitoring disease activity and (2) Validate the ability of the EST EBP to monitor therapeutic efficacy in 1-hour sampling time. The investigators supportive Preliminary Data demonstrate the feasibility of using ESTs in both children and adults with EoE to measure disease activity (esophageal inflammation) in an overnight (12-hour) test, and shorter time periods, currently performed before a scheduled endoscopy with biopsy. In this project, The investigators propose to shorten this time frame to a 1-hour test, a clinically relevant time point that will markedly facilitate its use and potential impact in the outpatient clinic setting.

Public Health Relevance/Impacts: At least four major impacts should result from these studies:

(1) Identification of an EBP will permit monitoring of esophageal inflammation in EoE; (2) the EBP will be relevant to following disease progression, treatment responses, management and pathogenesis of EoE, (3) validation of the EST EBP will enable development of rapid and inexpensive assays to follow treatment responses, thus reducing the number of follow-up endoscopies with biopsy that are currently performed, and (4) provide a device to monitor EoE disease activity where endoscopy with biopsy may not be available or affordable.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing esophagogastroduodenoscopy (EGD) at Children's Hospital Colorado, or
* Patients from a participating site in whom an inflammatory GI disease is suspected.
* Patients with symptoms of:

  1. abdominal pain,
  2. vomiting,
  3. growth delay, or
  4. malabsorption for which an etiology has not been determined.
* Patients with chronic eosinophilic esophagitis (EoE) in whom symptoms suggest ongoing inflammation.

Exclusion Criteria:

* Patients suffering from bleeding diathesis, or any other comorbid condition which their doctor feels may put them at additional risk.
* Patients with a family history of connective tissue disease.
* Patients undergoing a therapeutic endoscopy (such as dilatation, sclerotherapy, variceal banding).
* Patients with a history of:

  1. esophageal stricture, or
  2. surgery such as fundoplication, or
  3. allergy to gelatin, or
  4. inability to swallow pills.

Ages: 7 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Any pediatric or adult patient undergoing a clinically indicated endoscopy with biopsy at a participating site may be recruited. (initial cohort)
Sampling Method: Non-Probability Sample
Enrollment: 440 (Estimated)
Dates: Start 2009-01; Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Association of biomarker levels in biopsy tissue with pathological findings (eosinophil counts) | 12 weeks

SECONDARY OUTCOMES:
Correlation for the level of each biomarker between EST and tissue biopsy samples | 12 weeks

OTHER OUTCOMES:
Ability of an individual biomarker (or combination of biomarkers) to differentiate mucosal biopsy EBP sample obtained before and after treatment | 12 weeks
Ability of an individual biomarker (or combination of biomarkers) to differentiate post-treatment mucosal biopsy EBP sample from normal control | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Glenn T Furuta, MD, Principal Investigator — Children's Hospital Colorado
Locations (6):
- United States (6):
  - Children's Hospital Colorado, Aurora, Colorado
  - University of Colorado Hospital, Aurora, Colorado
  - Northwestern University, Chicago, Illinois
  - Lurie Children's Hospital, Chicago, Illinois
  - OSF St Francis Medical Center, Peoria, Illinois
  - Indiana University, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Furuta GT, Kagalwalla AF, Lee JJ, Alumkal P, Maybruck BT, Fillon S, Masterson JC, Ochkur S, Protheroe C, Moore W, Pan Z, Amsden K, Robinson Z, Capocelli K, Mukkada V, Atkins D, Fleischer D, Hosford L, Kwatia MA, Schroeder S, Kelly C, Lovell M, Melin-Aldana H, Ackerman SJ. The oesophageal string test: a novel, minimally invasive method measures mucosal inflammation in eosinophilic oesophagitis. Gut. 2013 Oct;62(10):1395-405. doi: 10.1136/gutjnl-2012-303171. Epub 2012 Aug 15. PMID 22895393
- [Background] Ackerman SJ, Kagalwalla AF, Hirano I, Gonsalves N, Katcher PM, Gupta S, Wechsler JB, Grozdanovic M, Pan Z, Masterson JC, Du J, Fantus RJ, Alumkal P, Lee JJ, Ochkur S, Ahmed F, Capocelli K, Melin-Aldana H, Biette K, Dubner A, Amsden K, Keeley K, Sulkowski M, Zalewski A, Atkins D, Furuta GT. One-Hour Esophageal String Test: A Nonendoscopic Minimally Invasive Test That Accurately Detects Disease Activity in Eosinophilic Esophagitis. Am J Gastroenterol. 2019 Oct;114(10):1614-1625. doi: 10.14309/ajg.0000000000000371. PMID 31567192